CLINICAL TRIAL: NCT04917549
Title: Prevalence of Oral Lesions in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, principal invistigator, Kafrelsheikh University
Other Study IDs: KD/04/20
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Oral Lesions; COVID-19; Angiotensin-converting Enzyme 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with COVID-19
  Interventions: Other: detection of oral lesions

INTERVENTIONS:
Other: detection of oral lesions — oral lesions in patient diagnosed with COVID-19

SUMMARY:
Recently, a new coronavirus disease 2019 (COVID-19) has appeared and caused an unprecedented pandemic which is considered as an urgent threat to health authorities worldwide. Several symptoms are observed which are fever, cough, shortness of breath, headache, runny nose, muscle pain, fatigue, arthralgia, sputum production, conjunctivitis, diarrhea. Susceptibility, genetics, systematic diseases, population, gender, and age are crucial considerations for the onset and progression of the viral infection. The patients suffering from asthma or pulmonary deficiency are at high risk of mortality. A metallopeptidase, angiotensin-converting enzyme 2 (ACE2) is considered as the functional receptor for SARS-CoV-2 and it was isolated from a COVID-19 patient. ACE2 was recognized in type I and type II alveolar epithelial cells in both nasal and oral mucosa, in the nasopharynx, in the smooth muscle cells and endothelium of vessels in the stomach and the skin, distinctly in the basal cell layer of the epidermis extending to the basal cell layer of hair follicles, and in the basal layer of the non-keratinizing squamous epithelium. In order to study the possible routes of SARS-CoV-2 infection on the oral mucosa, we investigated whether oral lesions mainly affect the tongue mucosa due to higher ACE2-expressing cell composition and proportion more than that in other oral tissues. Moreover, appearance of oral lesions were as a result of SARS-CoV-2 infection or as a side effect of certain drugs for COVID-19 treatment was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years.
* laboratory-confirmed COVID-19 infection (reverse transcription-polymerase chain reaction, RT-PCR).

Exclusion Criteria:

* patients without a laboratory-confirmed diagnosis of COVID-19 infection.
* patients with olfactory or gustatory dysfunctions before the epidemic.
* patients with some malignant neoplasms.
* patients with neurodegenerative disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All data was taken for each patient on the admission and during the hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
site of mucosa affected by oral lesions | 1 month
  Number and site of oral lesions that affect the oral cavity

SECONDARY OUTCOMES:
treatment of the patients | 1 month
  the correlation between the medications and the oral lesions

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Dalia Rasheed Issa, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The data are available upon request from the authors